CLINICAL TRIAL: NCT04409821
Title: COVID-19 Caregiver Emotional Support
Brief Title: Tele-based Psychological Emotional Support for Informal CARegivers of COVID-19 Patients in Intensive Care
Acronym: CO-CarES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Annika von Heymann, Postdoc, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: P-2020-544; 0216-00030B (Other Grant/Funding Number: Independent Research Fund Denmark)
Record Dates: First submitted 2020-05-22; First posted 2020-06-01 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Posttraumatic Stress Disorder; Prolonged Grief Disorder; COVID
Keywords: Informal caregiver; COVID-19
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Prolonged Grief Disorder; COVID-19

STUDY DESIGN:
Intervention Model Description: Feasibility study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tele-delivered psychological intervention (Experimental): Weekly tele-delivered psychological intervention
  Interventions: Behavioral: Tele-delivered psychological intervention

INTERVENTIONS:
Behavioral: Tele-delivered psychological intervention — The intervention consists of two (or one, if preferred by caregivers) weekly tele-sessions during the ICU stay, lasting up to 30 minutes, and two sessions in the month after discharge from or death in the ICU. Sessions will be conducted via phone-calls or video-conferencing. Therapists will 1) validate caregivers' subjective experience, 2) normalize and psychoeducate about emotional reactions, and 3) offer emotion regulation drawing on contemporary cognitive treatment packages of decentering, acceptance and emotion tolerance. Sessions for bereaved caregivers will include psycho-education about grief, assessment of risk for adverse outcomes and information about available support, if needed. The intervention will be performed based on an intervention manual. The content of the intervention will be continually adapted and tailored to the needs of the participating caregivers by involving all caregivers in co-creating the intervention trough brief post-session interviews.

SUMMARY:
The experience of a loved one's stay in a COVID-19 intensive care unit (ICU), either intubated or on respiratory support, forces family caregivers (hereafter 'caregivers') to face core existential fears, such as uncertainty and death. It also poses a serious threat to basic human needs for autonomy, competence, and relatedness, as family caregivers have no control over the illness, and limited prior competence in dealing with critical illness. COVID-19 likely aggravates this experience, as social distancing cuts caregivers off from visiting patients in the ICU, from using their usual social supportive network and the threat of infection extends to caregivers themselves, their children and family. Combined, these extreme circumstances put caregivers in emotional turmoil and in need of psychological support and assistance in managing difficult emotions. ICU caregivers are at risk of developing clinically relevant symptoms of anxiety or posttraumatic stress. During the patient's ICU stay, caregivers experience peri-traumatic distress, such as helplessness, grief, frustration and anger, that may predict later posttraumatic stress disorder (PTSD). Symptoms of anxiety and PTSD may last for months to years after the patient's discharge. Further, caregivers of patients who die in an ICU may be at greater risk of prolonged grief disorder. Supportive interventions may reduce psychological late effects in ICU caregivers, but the primary focus of the majority of interventions has been on communication or surrogate decision making. The CO-CarES study aims to develop and test the feasibility of a tele-delivered psychological intervention to enable caregivers of ICU patients with COVID-19 to better endure the overwhelming uncertainty and emotional strain and reduce the risk of posttraumatic stress and prolonged grief. The study hypothesizes that providing psychological intervention during and after the patients' hospitalization, can decrease peri-traumatic distress during ICU hospitalization and decrease risk of post-traumatic stress, anxiety, depression and perceived stress following discharge, as well as prolonged grief in bereavement. A secondary hypothesis is that changes in emotion regulation mediate effects of the intervention on long-term psychological outcomes.

ELIGIBILITY:
Inclusion Criteria:

* close relatives or friends of a patient hospitalized in an intensive care or intermediary care wards with COVID-19
* capable of completing online questionnaires
* speak Danish sufficiently for a therapeutic dialogue
* provide informed consent

Exclusion Criteria:

* suffering from a severe psychiatric disorder (such as schizophrenia) or in ongoing psychotherapeutic treatment for a psychiatric disorder (such as major depression generalized anxiety disorder or others), that cannot be paused
* unable to complete verbal phone- or videoconferencing calls
* unable to complete electronic questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-05-29 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | At inclusion
  Rate of consent among informed eligible participants
Completion rate | During and post-intervention (1 month)
  Rates of completion of intervention sessions among participants
Peri-traumatic distress inventory (negative emotions) | Pre-post intervention (1 month after discharge/death)
  Symptoms of peri-traumatic distress, min. score 0, max score 24, higher score corresponds to worse distress
Impact of Events Scale (6 item) | 1 month post intervention
  Posttraumatic stress, min. score 6, max score 24, higher score corresponds to worse distress
Impact of Events Scale (6 item) | 6 months post intervention
  Posttraumatic stress, min. score 6, max score 24, higher score corresponds to worse distress
Impact of Events Scale (6 item) | 12/13 months post intervention
  Posttraumatic stress, min. score 6, max score 24, higher score corresponds to worse distress

SECONDARY OUTCOMES:
Prolonged Grief-13-scale | 6 and 13 months
  Prolonged Grief, scored according to diagnostic criteria for prolonged grief disorder
PROMIS Depression (8 item scale) | Baseline to 1, 6, and 12/13 months
  Symptoms of depression, min. score 8, max score 40, higher score corresponds to worse symptoms
PROMIS Anxiety (8 item scale) | Baseline to 1, 6, and 12/13 months
  Symptoms of anxiety, min. score 8, max score 40, higher score corresponds to worse symptoms
Perceived Stress Scale (4 item) | Baseline to 1, 6, and 12/13 months
  Perceived stress, min. score 0, max score 16, higher score corresponds to worse stress

OTHER OUTCOMES:
Short Penn State Worry Questionnaire (3 items) | Baseline to 1, 6, and 12/13 months
  Worry, min. score 3, max score 15, higher score corresponds to greater worry
Brooding subscale of Ruminative Responses Scale | Baseline to 1, 6, and 12/13 months
  Brooding, min. score 5, max score 20, higher score corresponds to greater brooding/rumination
Intolerance of uncertainty Scale (2 item) | Baseline to 1, 6, and 12/13 months
  Intolerance of uncertainty, min score 2, max score 8, greater score indicates greater uncertainty intolerance

CONTACTS AND LOCATIONS:
Overall Officials: Annika von Heymann, PhD, Principal Investigator — Rigshospitalet, Denmark
Locations (6):
- Denmark (6):
  - Skejby Hospital, Aarhus
  - Rigshospitalet, Copenhagen
  - Hospitalsenheden Vest, Horsens, Horsens
  - Hvidovre Hospital, Hvidovre
  - Sygehus Lillebælt, Kolding, Kolding
  - Odense University Hospital, Odense

IPD SHARING:
Plan to Share IPD: No